CLINICAL TRIAL: NCT03227146
Title: A Phase IIb, Prospective, Intra-patient Randomised Controlled, Multicentre Study to Evaluate the Safety and Efficacy of an Autologous Bio-engineered Dermo-epidermal Skin Substitute (EHSG-KF) for the Treatment of Partial Deep Dermal and Full Thickness Burns in Adults and Adolescents in Comparison to Autologous Split-thickness Skin Grafts (STSG)
Brief Title: Study With an Autologous Dermo-epidermal Skin Substitute for the Treatment of Burns in Adults and Adolescents
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CUTISS AG (Industry)
Collaborators: Wyss Zurich (Unknown); Julius Clinical (Industry); Sintesi Research Srl (Industry); University Hospital, Zürich (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBRU-dS-BA-PIIb; NL62252.000.17; CS2/1421 (Other: Ethics NL; Ethics IT)
Record Dates: First submitted 2017-07-07; First posted 2017-07-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-01

CONDITIONS: Burns
Keywords: Burns; Scar; Skin; Wound healing; Tissue Engineering; Dermis; Epidermis; Thermal Injuries
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Option 1 (Other): Location A is the experimental area and Location B is the control area.
  Interventions: Biological: EHSG-KF; Biological: STSG
- Option 2 (Other): Location A is the control area and Location B is the experimental area.
  Interventions: Biological: EHSG-KF; Biological: STSG

INTERVENTIONS:
Biological: EHSG-KF — Transplantation of autologous dermo-epidermal skin substitute EHSG-KF to the experimental area
  Other Names: denovoSkin
Biological: STSG — Transplantation of autologous split-thickness skin graft to the control area
  Other Names: Split-thickness skin graft

SUMMARY:
This phase IIb trial aims to evaluate the efficacy and safety of EHSG-KF (synonym denovoSkin) in comparison to meshed STSG in adults and adolescents with partial deep dermal and full thickness burns.

DETAILED DESCRIPTION:
This multicentre phase IIb clinical trial will target adults and adolescents with severe burns to elucidate the benefit of a tissue-engineered autologous skin substitute for the patient group with the highest mortality rates. Particular emphasis, apart from safety, will be placed on efficacy, including the ratio of covered surface area to harvested surface area and scar quality, in comparison to meshed STSG.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥12 years of age
* Deep partial thickness and/or full thickness burns requiring surgical wound coverage
* Expected that ≥90 cm2 of wound (not counting the head and neck area for study patients in The Netherlands) will remain open at 4 weeks post burn despite proceeding with treatment in accordance with the standard of care. >20% TBSA burns can be taken as guideline, but TBSA is not an inclusion criterion.
* Signed Informed consent

Exclusion Criteria:

* Patients tested positive for HBV, HCV, syphilis or HIV
* Patients with known underlying or concomitant medical conditions that may interfere with normal wound healing (e.g. systemic skin and connective tissue diseases, any kind of congenital defect of metabolism including insulin-dependent diabetes mellitus, Cushing syndrome or disease, scurvy, chronic hypothyroidism, congenital or acquired immunosuppressive condition, chronic renal failure, or chronic hepatic dysfunction (Child-Pugh class B or C), severe malnutrition, or other concomitant illness which, in the opinion of the Investigator, has the potential to significantly delay wound healing)
* Severe drug and alcohol abuse
* Pre-existing coagulation disorders as defined by INR outside its normal value, PTT >ULN and fibrinogen <LLN prior to the current hospital admission and / or at the Investigator's discretion
* Patients with known allergies to amphotericin B, gentamicin, penicillin, streptomycin, or bovine collagen
* Previous enrolment of the patient into the current phase II study
* Participation of the patient in another study with conflicting endpoints within 30 days preceding and during the present study
* Patients expected not to comply with the study protocol (including patients with severe cognitive dysfunction/impairment and severe psychiatric disorders)
* Pregnant or breast feeding females
* Intention to become pregnant during the clinical course of the study (12 months)
* Wounds in the head and neck area as study target area (only applicable for study patients in The Netherlands)
* Enrolment of the Investigator, his/her family members, employees and other dependent persons

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of EHSG-KF in comparison to meshed STSG based on ratio of covered surface | 4 weeks post grafting
  Efficacy of EHSG-KF in comparison to meshed STSG based on ratio of covered surface area to biopsy site/donor site surface area

SECONDARY OUTCOMES:
Safety of EHSG-KF in comparison to meshed STSG based on clinical signs of infection | 4-11 days post grafting and 21 +/-2 days post grafting
  Evaluation of clinical signs of infection at experimental area and control area
Safety of EHSG-KF in comparison to meshed STSG based on microbiological signs of infection | 4-11 days post grafting and 21 +/-2 days post grafting
  Evaluation of microbiologic signs of infection at experimental area and control area
Efficacy of EHSG-KF in comparison to meshed STSG based on evaluation of scar quality by measurement of the elasticity using Cutometer(R) | 1 year +/-30 days post grafting
  Assessment of elasticity of experimental area and control area using Cutometer(R)
Efficacy of EHSG-KF in comparison to meshed STSG based on evaluation of scar quality by assessment of General scar quality using POSAS assessment tool | 1 year +/-30 days post grafting
  Assessment of general scar Quality of experimental area and control area using POSAS assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Schiestl, Prof., Study Chair — University Children's Hospital, Zurich
Locations (6):
- Italy (2):
  - Chirurgia Plastica e Centro Grandi Ustioni Azienda Ospedaliera di Rilievo Nazionale A. Cardarelli, Napoli
  - Unità di Chirurgia Plastica e Ustioni Ospedale Santobono, Napoli
- Netherlands (2):
  - Rode Kruis Ziekenhuis, Beverwijk
  - Maasstad Ziekenhuis, Rotterdam
- Switzerland (2):
  - University Children's Hospital Zurich, Zurich, Canton of Zurich
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meuli M, Schiestl C, Hartmann-Fritsch F, Middelkoop E, Kim BS, Neuhaus K, Plock JA, Rittirsch D, van der Vlies CH, Azzena B, Marino D, Mujynya K, Farkas M, Bressan J, Reichmann E, Bottcher-Haberzeth S. Safety and efficacy of bio-engineered, autologous dermo-epidermal skin grafts in adolescent and adult burn patients: 1-year results of a prospective, randomized, controlled, multicenter phase IIB clinical trial. EClinicalMedicine. 2025 Nov 28;90:103665. doi: 10.1016/j.eclinm.2025.103665. eCollection 2025 Dec. PMID 41399471
- [Derived] Schiestl C, Neuhaus K, Meuli M, Farkas M, Hartmann-Fritsch F, Elrod J, Bressan J, Reichmann E, Bottcher-Haberzeth S. Long-Term Outcomes of a Cultured Autologous Dermo-Epidermal Skin Substitute in Children: 5-Year Results of a Phase I Clinical Trial. J Burn Care Res. 2025 Mar 4;46(2):326-334. doi: 10.1093/jbcr/irae150. PMID 39115183